CLINICAL TRIAL: NCT01282177
Title: Monitoring Seasonal and Pandemic Vaccine Safety and Effectiveness in Healthcare Providers:A Prospective Cohort Study
Brief Title: Influenza Vaccine Safety and Effectiveness in Healthcare Providers
Status: Completed | Type: Observational
Sponsor: Dalhousie University (Other)
Collaborators: PHAC/CIHR Influenza Research Network (Other Government)
Responsible Party: Principal Investigator, Shelly A. McNeil, Principal Investigator, Dalhousie University
Other Study IDs: 114142
Record Dates: First submitted 2011-01-07; First posted 2011-01-24 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Influenza
Keywords: surveillance, safety , tolerability , vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of this study is to provide ongoing assessment of the safety and effectiveness of seasonal and pandemic H1N1 vaccines in the prevention of ILI (influenza like illness), ILI-associated work absenteeism, and laboratory-confirmed influenza in a cohort of Canadian HCP (Health care providers). Given the uncertainties around the timing of the provision of seasonal influenza immunization to HCP for the 2009/10 influenza season, this study will focus on evaluation of safety and effectiveness of pandemic influenza immunization in Year 1 and evaluation of all recommended influenza vaccines in Years 2 and 3.

DETAILED DESCRIPTION:
Participants in Year 1 (2009/10) will be recruited beginning Oct. 1 through the end of the pandemic H1N1 influenza immunization campaign.

Participants will be followed from the day of vaccination until the end of the influenza season approximately Oct-April for each season.

At the initial visit, participants will have 1 tube of blood (10cc) collected at the time of enrolment to determine baseline antibody titres against pandemic H1N1 and the influenza strains in the past and current year's seasonal influenza vaccines.

Participants will receive automated email reminders with links to follow-up web-based questionnaires at weekly intervals following the completion of the baseline survey and until the end of the influenza season.

If a participant reports a respiratory illness, they will receive a follow-up questionnaire asking details of the illness including the occurrence of respiratory illness and associated symptoms, contact with patients or household members that had respiratory illness, respiratory symptom-related healthcare utilization, prescription or over-the-counter products used for treatment of the respiratory illness, and number of days of work missed due to respiratory illness or worked with symptomatic respiratory tract infection. An email will be sent to each participant every Monday morning during the season reminding the participant to complete their weekly diary and report and send in their nasal swab if they have symptoms of an acute respiratory illness.

At the initial visit participants will be taught how to collect their nasal swab and will practice doing their own swab in the presence of the study nurse/research associate. Participants will be instructed to collect a nasal swab and return the swabs as soon as possible after onset of ILI or respiratory illness (target < 48h after onset). Participants will be asked to collect the swab if they develop symptoms compatible with a viral respiratory tract infection (fever without an apparent source OR new symptoms with at least 2 of the following -cough, runny/stuffy nose, sneezing, sore/scratchy throat, hoarseness, malaise, myalgia, headache, fatigue OR one local symptom (runny/stuffy nose, sneezing, sore/scratchy throat, hoarseness, cough) plus one systemic symptom (fever, malaise, myalgia, headache, fatigue). If they prefer, a nasopharyngeal swab will be collected by a member of the study team as soon as possible after the onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1)18-69 years old, inclusive, as of Sept. 1 on the year of enrolment; 2)understand the study, agree to its provisions, and give written informed consent to participate; 3)available for follow-up for at least 1 influenza season 4)have convenient access to a computer with internet access and basic skills for use of the internet; 5)employed full-or part -time (> 8 hours/week) in an acute care hospital (in any occupation) or, if a physician or midwife, working at least 8 hours per week in an acute care hospital.

Exclusion Criteria:

1. planning to spend more than two consecutive weeks outside of Canada during the winter study period (Oct. 15- Apr. 15);
2. received an immunoglobulin within 6 months of study entry;
3. planning to take leave from work for more than two consecutive weeks during the winter study period (e.g. maternity or medical leave);
4. participating in a trial that would result in receipt of an investigational medication during the study period

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of adult HCP will be offered the opportunity to participate in this surveillance study at Influenza vaccination clinics in their health care facility
Sampling Method: Non-Probability Sample
Enrollment: 1143 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of seasonal and pandemic influenza vaccine among a cohort of HCP | October to April each year
  Health care providers will receive automated email reminders with a link to report any changes in their health within 4 weeks of vaccination.

SECONDARY OUTCOMES:
To validate published ILI case definitions in a cohort of HCP | October to April each year
  A cohort of HCP will be asked via an automated email to report the presence of an upper respiratory illness and to self collect a nasal swab to be tested for influenza.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly A McNeil, MD, Principal Investigator — Dalhousie University; Allison McGeer, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Anne McCarthy, MD, Principal Investigator — The Ottawa Hospital; Mark Loeb, MD, Principal Investigator — Hamilton Health Sciences Center; Grant Stiver, MD, Principal Investigator — Vancouver General Hospital; Brenda Coleman, MD, Principal Investigator — MOUNT SINAI HOSPITAL